CLINICAL TRIAL: NCT01952626
Title: Prevention of Intrathecal Morphine Induced Pruritus: Comparison of Ondansetron and Palonosetron
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Younghoon Jeon, Associate professor, Kyungpook National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KNUH 2013-03-032-001
Record Dates: First submitted 2013-06-11; First posted 2013-09-30 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Morphine Adverse Reaction
Keywords: intrathecal; morphine; ondansetron; palonosetron; pruritus
MeSH Terms: conditions — Pruritus | interventions — Ondansetron; Palonosetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ondansetron (Active Comparator): Intravenous administration of ondansetron 4mg 15 minutes before spinal anesthesia
  Interventions: Drug: Ondansetron
- palonosetron (Experimental): Intravenous administration of palonosetron 0.075mg 15 minutes before spinal anesthesia
  Interventions: Drug: Palonosetron

INTERVENTIONS:
Drug: Ondansetron — intravenous injection
  Other Names: zofran
  Arms: ondansetron
Drug: Palonosetron — intravenous injection
  Other Names: aloxi
  Arms: palonosetron

SUMMARY:
Intrathecal administration of morphine is often used for control of postoperative pain. However, pruritus is one of the most common side effects of intrathecal morphine . Specific serotonin receptor antagonists could be an effective prophylactic treatment of neuraxial opioid-induced pruritus. It was reported that palonosetron is more effective than ondansetron for prevention of postoperative nausea and vomiting. Therefore, the investigators evaluated the efficacy of prophylactic administration of ondansetron and palonosetron for the prevention of intrathecal morphine-induced pruritus.

DETAILED DESCRIPTION:
Intrathecal administration of morphine is often used for relief of postoperative pain. However, pruritus is one of the most common side effects associated with intrathecal morphine. Specific serotonin receptor antagonists such as ondansetron could be an effective prophylactic treatment of neuraxial opioid-induced pruritus. It was reported that palonosetron is more effective than ondansetron for prevention of postoperative nausea and vomiting. Therefore, the investigators evaluated the efficacy of prophylactic administration of ondansetron and palonosetron for the prevention of intrathecal morphine-induced pruritus.

ELIGIBILITY:
Inclusion Criteria:

* 19-70 years,
* American Society of Anesthesiology physical status 1 and 2
* Scheduled for elective urologic surgery under spinal anesthesia.

Exclusion Criteria:

* Patients with cardiac and psychological problems.
* Patients who take sedatives or narcotics.
* Patient who have allergy to study drugs.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Incidence of pruritus | 24 hours after spinal anesthesia
  record of the incidence of pruritus after spinal anesthsia

CONTACTS AND LOCATIONS:
Overall Officials: Younghoon Jeon, Dr, Principal Investigator — Kyungpook National University Hopsital
Locations (1):
- Kyungpook National Hospital, Daegu, South Korea